CLINICAL TRIAL: NCT04594018
Title: National, Multicentre, Randomized, Double-blind, Double-dummy Phase III Clinical Trial to Evaluate the Efficacy and Safety of Finlândia Hair Lotion Association in the Treatment of Androgenetic Alopecia.
Brief Title: Efficacy and Safety of Finlândia Hair Lotion Association on Androgenetic Alopecia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS2119 - FINLÂNDIA
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia
Keywords: androgenetic alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Finasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FINLÂNDIA (Experimental): The study is double-dummy. The patient must take 1 pill and apply hair lotion as follow:
  1 tablet finasteride placebo, oral, once a day.
  1 mL Finlândia hair lotion, topical, twice a day.
  Interventions: Drug: Finlândia Association + finasteride placebo
- Minoxidil + finasteride (Active Comparator): The study is double-dummy. The patient must take 1 pill and apply hair lotion as follow:
  1 tablet finasteride, oral, once a day.
  1 mL minoxidil hair lotion, topical, twice a day.
  Interventions: Drug: Minoxidil + finasteride

INTERVENTIONS:
Drug: Finlândia Association + finasteride placebo — Finlândia association hair lotion + finasteride placebo
  Arms: FINLÂNDIA
Drug: Minoxidil + finasteride — Minoxidil hair lotion + Finasteride 1 mg
  Arms: Minoxidil + finasteride

SUMMARY:
The purpose of this study is to evaluate the efficacy of Finlândia hair lotion association in the treatment of androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Men aged 18 years or over and less than or equal to 60 years with a diagnosis of Androgenetic Alopecia grades IIIv to IV in the modified Norwood-Hamilton classification, who have been using minoxidil 5% for at least 3 months and willing to maintain the same style, approximate length and hair color throughout the test.

Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* History of alcohol and/or substance abuse within 2 years;
* Participants with other concomitant dermatological diseases on the scalp, except for mild seborrhoea dermatitis;
* Participants with a history of surgical treatment for hair loss or shaved scalp;
* Participants who used shampoo or topical solution containing ketoconazole, tar, selenium, threonine or steroids in the last 2 weeks;
* Participants who used 5α reductase inhibitors, such as finasteride and dutasteride, in the last 12 months;
* Participants using testosterone replacement therapy (TRT) or using testosterone-containing gel;
* Participants who used micro-infusion of medications on the skin (MMP), microneedling or intradermotherapy on the scalp in the last 3 months;
* Participants who have undergone radiation treatment for the scalp or chemotherapy in the past year;
* Participants with diseases that can affect hair growth;
* Participants with a current medical history of cancer and / or cancer treatment in the last 5 years;

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hair density. | 6 months
  Digital phototrichogram evaluation of vertex area regarding the change from baseline in number of hairs after 6 months of treatment compared to baseline.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto Da Pele, Osasco, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No